CLINICAL TRIAL: NCT05321238
Title: The Role of Agency and Threat-Immediacy in Interactive Digital Narrative Fear Appeals for the Prevention of Excessive Alcohol Use: Randomized Controlled Trial
Brief Title: The Role of Agency and Threat-Immediacy in Interactive Digital Narrative Fear Appeals
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Tilburg University (Other)
Responsible Party: Principal Investigator, Hendrik Engelbrecht, Principal Investigator, Tilburg University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 2020.141
Record Dates: First submitted 2022-04-01; First posted 2022-04-11 (Actual); Last update posted 2022-04-22 (Actual); Status verified 2022-04

CONDITIONS: Excessive Drinking
Keywords: agency; fear appeal; alcohol; narrative
MeSH Terms: conditions — Narration

STUDY DESIGN:
Who Masked: Participant
Masking Description: Participants were not aware which arm of the study they were enrolled in.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- High agency and immediate threat (Experimental): Participants were asked to make decisions within the interactive digital narrative and were presented with acute alcohol poisoning of the main character in the story.
  Interventions: Other: High agency and immediate threat
- High agency and distant threat (Experimental): Participants were asked to make decisions within the interactive digital narrative and were presented with multiple organ failure after years of alcohol consumption of the main character in the story.
  Interventions: Other: High agency and distant threat
- Low agency and immediate threat (Experimental): Participants were presented with a fixed (passive) narrative without decisions and were presented with acute alcohol poisoning of the main character in the story.
  Interventions: Other: Low agency and immediate threat
- Low agency and distant threat (Experimental): Participants were presented with a fixed (passive) narrative without decisions and were presented with multiple organ failure after years of alcohol consumption of the main character in the story.
  Interventions: Other: Low agency and distant threat

INTERVENTIONS:
Other: High agency and immediate threat — Participants were asked to make several decisions for the main character in the interactive digital narrative that related to drinking / turning down alcoholic drinks.The decisions made lead to a ending consistent with the decisions of the participant. In the story presented, a character dies from acute alcohol poisoning after ingesting too much alcohol in a short period of time.
  Arms: High agency and immediate threat
Other: High agency and distant threat — Participants were asked to make several decisions for the main character in the interactive digital narrative that related to drinking / turning down alcoholic drinks.The decisions made lead to a ending consistent with the decisions of the participant. In the story presented, a character dies from multiple organ failure after ingesting too much alcohol over a long period of time.
  Arms: High agency and distant threat
Other: Low agency and immediate threat — Participants were asked to read a narrative in which the main character turns down alcoholic drinks at a party. The participants can not influence the decisions of the main character and only consume the narrative passively.The decisions made lead to a ending consistent with the decisions of the participant. In the story presented, a character dies from acute alcohol poisoning after ingesting too much alcohol in a short period of time.
  Arms: Low agency and immediate threat
Other: Low agency and distant threat — Participants were asked to read a narrative in which the main character turns down alcoholic drinks at a party. The participants can not influence the decisions of the main character and only consume the narrative passively.The decisions made lead to a ending consistent with the decisions of the participant. In the story presented, a character dies from multiple organ failure after ingesting too much alcohol over a long period of time.
  Arms: Low agency and distant threat

SUMMARY:
Aims:

The first aim of the study was to assess the effect of agency, i.e. the perception of making meaningful decisions, in an interactive digital narrative fear appeal on self-efficacy beliefs concerning the ability to reduce alcohol intake among college students. Second, we assessed whether the communicated timeframe (short-term / long-term) of the threat presented in the narrative moderates the effect of agency on self-efficacy. Lastly, to validate the effect of the intervention on behavioural outcomes we assesed whether self-efficacy has an effect on behavioural intention measures.

The study was a 2 (agency: low / high) x 2 (time-frame: immediate / distant) between-subjects online experiment.

ELIGIBILITY:
Inclusion Criteria:

* above 18 years of age
* 480 seconds survey completion time
* both attention checks relating to narrative content passed
* correctly identified their experimental condition in the manipulation check
* did not choose to 'drink an alcoholic drink' for all decisions in the interactive narrative
* did not show signs of alcohol abuse

Exclusion Criteria:

* under the age of 18
* completed the questionnaire in an unreasonably short amount of time
* they failed one of the two attention checks
* failed the manipulation check asking them to recall whether they were presented with short- or long-term (high / low immediacy) consequences of excessive drinking
* chose an alcoholic drink for all decision points
* showed signs of alcohol dependence as measured above 15 on the Brief Young Adult Alcohol Consequences Questionnaire (B-YAACQ)

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 178 (Actual)
Dates: Start 2020-11-26 (Actual); Primary Completion 2020-12-18 (Actual); Study Completion 2020-12-18 (Actual)

PRIMARY OUTCOMES:
Perceived self-efficacy | During the lab session
  Three items answered on 7-point Likert scales (ranging from 'Strongly Disagree' to 'Strongly Agree'):
  1. I am able to limit my alcohol intake to low amounts.
  2. It is easy for me to limit my alcohol intake to low amounts.
  3. I can limit my alcohol intake to low amounts.
Behavioural intention | During the lab session
  Four items answered on 7-point Likert scales (ranging from 'Strongly Disagree' to 'Strongly Agree'):
  1. I intend to limit my alcohol intake to low amounts.
  2. I intend to limit my alcohol intake to low amounts on special occasions.
  3. I intend to limit my alcohol intake to low amounts when being with friends.
  4. I intend to limit my alcohol intake to low amounts when I am by myself.

OTHER OUTCOMES:
Perceived Agency | During the lab session
  Five items Items were measured on 7-point Likert scales from 'Strongly Disagree' to 'Strongly Agree'. For example, 'I felt that the actions I took were meaningful within the context of the story'.
Fear | During the lab session
  Six items were scored on 7-point Likert scales from 'Not at all' to 'Very much'. The items ask participants about the intensity of affective response towards the message, for example, 'How much did this message make you feel frightened?'.
Perceived Severity, Susceptability and Response-Efficacy | During the lab session
  Severity, susceptibility and response-efficacy items were measured with three items each on 7-point Likert scales from 'Strongly Disagree' to 'Strongly Agree'.
Symptoms of Alcohol Abuse | During the lab session
  We measured the consequences of alcohol related behavior indicating dependence. One example of an item is 'My drinking has gotten me into sexual situations I later regretted.'. The brief young adult alcohol consequences questionnaire (BYAACQ) consists of 24 statements that are scored with binary yes / no answers. A score above 15 positive answers indicates alcohol dependence. The scale was developed by (Kahler et al., 2008).
Drinking Frequency | During the lab session
  Frequency was measured by asking participants how often they 'drink alcohol in excess' and was measured on a 7-point Likert scale ranging from 'Never' to 'Very Frequently'.
Perceived Control | During the lab session
  Perceived control was measured by two items asking participants whether or not they can 'control' and 'stop' drinking alcohol whenever they want. These two items were measured on 7-point Likert scales ranging from 'Strongly Disagree' to 'Strongly Agree'.
Behavioural inhibition | During the lab session
  The items to measures disinhibition were taken over unchanged from the scale by Lee & Shinn (2011), but altered from 9-point to 7-point Likert scales ranging from 'Strongly Disagree' to 'Strongly Agree'.

CONTACTS AND LOCATIONS:
Overall Officials: Hendrik Engelbrecht, Principal Investigator — Tilburg University
Locations (1):
- Tilburg University, Tilburg, North Brabant, Netherlands

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Engelbrecht H, van der Laan LN, van Enschot R, Krahmer E. The Role of Agency and Threat Immediacy in Interactive Digital Narrative Fear Appeals for the Prevention of Excessive Alcohol Use: Randomized Controlled Trial. JMIR Serious Games. 2022 Jun 13;10(2):e32218. doi: 10.2196/32218. PMID 35699976